CLINICAL TRIAL: NCT05526235
Title: Reducing the Psychosocial Impact of the Covid-19 Pandemic on Workers of Assisted Living Facilities
Brief Title: A Scalable Psychological Intervention to Reduce Psychological Distress Among Workers of Assisted Living Facilities
Acronym: REPICAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: VU University of Amsterdam (Other); Universidad Autonoma de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202114
Record Dates: First submitted 2022-07-21; First posted 2022-09-02 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Depression; Anxiety; Psychological Distress
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Psychological First Aid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepped-care program (Step 1: DWM; Step 2: PM+) (Experimental): The treatment group will first receive Psychological First Aid (PFA). PFA consists of a 15-min call that assess the immediate concerns and needs of an individual in order to connect individuals to help and resources.
  Afterwards participants will receive the stepped-care program consisting of Doing What Matters (DWM) (step 1) and Problem Management Plus (PM+) (step 2). Step 2 will only be provided if the participant still has elevated levels of psychological distress (i.e. during the second quantitative assessment at 2 weeks after DWM).
  Participants will also be allowed to continue with their mental health interventions (CAU), as long as they meet eligibility criteria.
  Interventions:
  Behavioral: Doing What Matters (DWM) Behavioral: Problem Management Plus (PM+) Behavioral: Psychological First Aid (PFA)
  Interventions: Behavioral: Doing What Matters (DWM); Behavioral: Problem Management Plus (PM+); Behavioral: Psychological First Aid (PFA)
- Psychological First Aid (PFA) (Active Comparator): Participants allocated to the control arm will also receive PFA. Participants will also be allowed to continue with their mental health interventions (CAU), as long as they meet eligibility criteria.
  Intervention: Behavioral: Psychological First Aid (PFA)
  Interventions: Behavioral: Psychological First Aid (PFA)

INTERVENTIONS:
Behavioral: Doing What Matters (DWM) — The original DWM program consists of a self-help guide called 'Doing What Matters in Times of Stress', that is complemented with pre-recorded audio exercises. The audio material imparts key information about stress management and guides participants through individual exercises. Additionally, participants are guided by a briefly trained helper. In this study, DWM will be delivered as an online intervention. The DWM intervention, i.e. both the audio recordings and the self-help guide, has been adapted for use on a smartphone or other device with internet access. The format of DWM is innovative in that it seeks to ensure that key intervention components are delivered as intended through the use of pre-recorded audio, without the burden of extensive training and supervision. In the online application tool a new module is released every week so participants will be asked to go through the entire DWM intervention within 5 weeks with weekly guidance from a helper.
  Other Names: Doing What Matters in Times of Stress; Self Help Plus; DWM; SH+
  Arms: Stepped-care program (Step 1: DWM; Step 2: PM+)
Behavioral: Problem Management Plus (PM+) — PM+ is a new, brief, psychological intervention program based on cognitive behavioral therapy (CBT) techniques. The manual involves the following empirically supported elements: problem solving plus stress management, behavioral activation, facing fears, and accessing social support. Across the five 90-minute sessions participants may talk to trained non-professional. PM+ has four core features, and it is brief. In this study, the delivery mode of the PM+ intervention will be flexible, with remote delivery in phases of the pandemic when physical distancing rules apply. This is a future-oriented attempt towards a more holistic mental health care system that can flexibly switch between modes of delivery (e.g. remotely (e.g. Zoom) or face-to), depending on the needs and the specific containment measures that apply, and the specific preferences and needs of the participant.
  Other Names: PM+
  Arms: Stepped-care program (Step 1: DWM; Step 2: PM+)
Behavioral: Psychological First Aid (PFA) — PFA is a brief intervention consisting of a 15-min call that assess the immediate concerns and needs of an individual in order to connect individuals to help and resources.
  Other Names: PFA

SUMMARY:
The current study is a randomized controlled trial (RCT) that aims to evaluate the effectiveness of a stepped-care program (Doing What Matters [DWM] and Problem Management Plus [PM+]) in reducing anxiety and depression symptoms amongst long-term care workers (LTCWs), following changes in care due to the COVID-19 pandemic.

DETAILED DESCRIPTION:
Background: The COVID-19 pandemic has impacted the mental health of long-term care workers (LTCWs). This study combines two low-intensity psychological interventions developed by the World Health Organization (Doing What Matters [DWM] and Problem Management Plus [PM+]) into a stepped-care program for LTCWs.

Objective: To evaluate the implementation of a stepped-care program (DWM; PM+) amongst LTCWs following changes in care due to the COVID-19 pandemic in terms of mental distress, resilience and wellbeing.

Study design: A randomized controlled implementation trial with a single-blinded, parallel-group design.

Study population: Long-term care workers (including workers of assisted living facilities and home care) with self-reported elevated psychological distress.

Intervention-study: All participants (in both the treatment and the comparison group) will receive Psychological First Aid (PFA) and care as usual (CAU). In addition to PFA and CAU, the treatment group will receive the stepped-care intervention (DWM with or without PM+). The stepped-care intervention consists of DWM (step 1) and conditionally PM+ (step 2) if participants still meet criteria for psychological distress (Kessler Psychological Distress scale (K10) >15.9) 1 month after having received DWM.

Main study parameters/endpoints: Screening for inclusion and exclusion criteria will be interviewer-administered through phone calls. All assessments will be online and will take place at baseline, 2 weeks after having received DWM, 1 week after having received PM+ and 2 months after PM+. The main study parameter will be the decrease of anxiety and depressive symptoms from baseline to two-month follow-up, measured through the sum score of the Patient Health Questionnaire (PHQ-9) and General Anxiety Disorder-7 (GAD-7), i.e. the PHQ-Anxiety and Depression Score (PHQ-ADS).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* Having elevated levels of psychological distress (Kessler Psychological Distress Scale (K10) >15.9).
* Written/digital informed consent before entering the study.
* Being a worker in a long-term care facility or a home care worker in the community of Catalonia.

Exclusion Criteria:

* Having acute medical conditions (requiring hospitalization)
* Imminent suicide risk, or expressed acute needs, or protection risks that require immediate follow-up
* Having a severe mental disorder (e.g., psychotic disorders, substance-dependence)
* Having severe cognitive impairment (e.g., severe intellectual disability or dementia)
* Currently specialized psychological treatment (e.g., Eye movement desensitization and reprocessing, Cognitive behavioral therapy)
* In case of current psychotropic medication use, being on an unstable dose for at least 2 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS) | Change from baseline to 20 weeks
  The PHQ-ADS is a 16-item self-reported instrument that combines the nine-item Patient Health Questionnaire depression scale and seven-item Generalized Anxiety Disorder scale-as a composite measure of depression and anxiety. Respondents are asked how much each symptom has bothered them over the past 2 weeks, with response options of "not at all", "several days", "more than half the days", and "nearly every day", scored as 0, 1, 2, and 3. The scale can range from 0 to 48, with higher scores indicating higher levels of depression and anxiety symptomatology.

SECONDARY OUTCOMES:
Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS) | Change: Baseline, 6 weeks, and 12 weeks
  The PHQ-ADS is a 16-item self-reported instrument that combines the nine-item Patient Health Questionnaire depression scale and seven-item Generalized Anxiety Disorder scale-as a composite measure of depression and anxiety. Respondents are asked how much each symptom has bothered them over the past 2 weeks, with response options of "not at all", "several days", "more than half the days", and "nearly every day", scored as 0, 1, 2, and 3. The scale can range from 0 to 48, with higher scores indicating higher levels of depression and anxiety symptomatology.
Patient Health Questionnaire (PHQ-9) | Baseline, 6 weeks, 12 weeks, and 20 weeks
  The PHQ-9 is a 9-item self-reported instrument that measures depression symptoms. Respondents are asked how much each symptom has bothered them over the past 2 weeks, with response options of "not at all", "several days", "more than half the days", and "nearly every day", scored as 0, 1, 2, and 3. The scale can range from 0 to 27, with higher scores indicating higher levels of depression.
Generalized Anxiety Disorder (GAD-7) scale | Change: Baseline, 6 weeks, 12 weeks, and 20 weeks
  The GAD-7 is a 7-item self-reported instrument that measures anxiety symptoms. Respondents are asked how much each symptom has bothered them over the past 2 weeks, with response options of "not at all", "several days", "more than half the days", and "nearly every day", scored as 0, 1, 2, and 3. The scale can range from 0 to 21, with higher scores indicating higher levels of anxiety.
Posttraumatic Stress Disorder (PTSD) Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (PCL-5) - 8-item version | Change: Baseline, 6 weeks, 12 weeks, and 20 weeks
  The PCL-5 is a self-reported instrument that measures PTSD symptoms. Respondents are asked how much each symptom has bothered them over the past 4 weeks, with response options of "not at all", "a little bit", "moderately", "quite a bit", and "extremely". Items are rated on a 0-4 scale. The scale can range from 0 to 32 for the 8-item version, with higher scores indicating higher levels of PTSD symptoms.
EuroQol 5-dimensional descriptive system - 5-level version (EQ-5D-5L) | Baseline, 6 weeks, 12 weeks, and 20 weeks
  The EQ-5D-5L measures quality of life and consists of two parts, the EQ-5D and the EQ VAS. Part 1, the EQ-5D, rates the level of impairment across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The labels for the 5L followed the format "no problems," "slight problems," "moderate problems," "severe problems," and "unable to"/"extreme problems" for all dimensions. For mobility, the description of "confined to bed" has been changed to "unable to walk about.". Part 2, the EQ-VAS, is a visual analogue scale. The endpoints of the scale are called 'The best health you can imagine' and 'The worst health you can imagine' and the current health status of that day needs to be indicated, after which the number checked on the scale also needs to be written down. Higher scores indicate worst qualitive of life.
Client Service Receipt Inventory (CSRI) - adaptation | Change: Baseline, 6 weeks, 12 weeks, and 20 weeks
  The CSRI was developed for the collection of data on service utilization (e.g. use of health system, other services, time out of employment and other usual activities, need for informal care) and related characteristics of people with mental disorders, as the basis for calculating the costs of care for mental health cost-effectiveness research. The RESPOND-adapted version consists of a 13-item self-reported instrument that asks about the number and duration of contacts with healthcare professionals (physicians, mental health specialists, and nurses) in the past two months.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Maria Haro, MD,PhD, Principal Investigator — Fundació Sant Joan de Déu
Locations (1):
- Parc Sanitari Sant Joan de Déu, Sant Boi de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided